## **Study protocol**

Version 1, 2009-11-30

## Malmö Breast Tomosynthesis Screening Trial, MBTST

## **Principal investigator**

Sophia Zackrisson MD, PhD

Department of Translational Medicine, Diagnostic Radiology

Lund University and Skåne University Hospital Malmö

sophia.zackrisson@med.lu.se

## Synopsis

| Study title | Malmö Breast Tomosynthesis Screening Trial, MBTST |
|---|---|
| | http://www.clinicaltrials.gov/; NCT01091545 |
| Study phase | N/A |
| Background | Digital breast tomosynthesis, DBT (or 3D mammography) is a development of the currently used method in breast cancer screening, digital mammography, DM, that may increase the visibility of breast cancers and hence the detection. |
| Study setting | Within the population based screening programme in Malmö, Sweden. Skåne University Hospital Malmö, Unilabs Breast Centre. |
| Study design | Prospective, paired, one-armed study in a population-based screening program |
| Objectives | Primary objective: • to investigate the sensitivity and specificity of breast cancer detection with DBT compared to DM. |
| | Secondary objectives: - to investigate the biological characteristics of the cancers in the trial by |

| | mode of detection |
|---|---|
| | - to investigate the cost-effectiveness of DBT in screening |
| Study population | Inclusion criteria: a random selection of women aged 40-74 years invited to participate in mammography screening in Malmö |
| | Exclusion criteria: Pregnancy and/or women not understanding Swedish or English |
| Methods | Women will undergo both DBT in the medio-lateral oblique (MLO) |
| | projection and DM in MLO as well as cranio-caudal projection (CC). Reading of DBT and DM will be done independently. In addition, the DBT examination will be read together with the DM CC-view in order to assess the separate contribution of the DM CC-view. All studies will be double read. |
| | A two-year follow up and matching to the cancer registry will be performed to ascertain screening detected cancers and interval cancers. |
| Assessments | Women who are recalled for further assessment based on any method will be investigated according to so called triple assessment. |
| Statistical considerations | About 15,000 women are needed for this study in order to yield an 80% chance of getting a statistically significant outcome, i.e. detecting an increase in TPF and confirming that the FPF is within the acceptable limit of 20%. |
| Potential<br>benefit: | An improved breast cancer detection with DBT may increase the benefits of breast cancer screening and further contribute to reduced mortality in breast cancer. |